CLINICAL TRIAL: NCT05493618
Title: A Phase II Study of Pembrolizumab, Belantamab and Dexamethasone in Patients With Triple Class Refractory Multiple Myeloma.
Brief Title: Pembrolizumab, Belantamab and Dexamethasone in Refractory Multiple Myeloma.
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study Drug Unavailability
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro2022-0093; ISS 60989 (Other Grant/Funding Number: Merck)
Record Dates: First submitted 2022-08-05; First posted 2022-08-09 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Multiple Myeloma, Refractory
MeSH Terms: conditions — Multiple Myeloma | interventions — pembrolizumab; belantamab mafodotin; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: Safety lead-in Cohort: After the first 10 patients are enrolled, an independent safety review committee will meet to review adverse events and toxicity and determine whether the trial will continue to enroll.
  Phase 2 portion: The remainder of patients will be enrolled using a Simon's - 2 stage design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-arm, multi-institution (Experimental): Study Arm:
  Pembrolizumab 200 mg IV q3 weeks Belantamab 2.5 mg/kg IV q3 weeks. Dex 40 mg IV q3 weeks (20 mg if patient >75) Treatment will be administered on a 21-day cycle and will be continued until unacceptable toxicity or disease progression for up to 2 years (35 cycles)
  Interventions: Drug: Pembrolizumab; Drug: Belantamab mafodotin; Drug: Dexamethasone

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg IV q3 weeks until unacceptable toxicity or disease progression for up to 2 years (35 cycles).
  Other Names: Keytruda
Drug: Belantamab mafodotin — Belantamab 2.5 mg/kg IV q3 weeks until unacceptable toxicity or disease progression for up to 2 years (35 cycles).
  Other Names: Blenrep
Drug: Dexamethasone — Dexamethasone 40 mg IV q3 weeks (20 mg if patient >75) until unacceptable toxicity or disease progression for up to 2 years (35 cycles).
  Other Names: Decadron

SUMMARY:
This is a single arm, multi-institution (1) Hackensack Meridian Health at Hackensack, New Jersey (NJ) (2) Jersey Shore Medical Center, Neptune, NJ and (3) Georgetown/Lombardi Cancer Center) phase II study of the combination of pembrolizumab, belantamab, and dexamethasone in patients with triple class refractory multiple myeloma.

DETAILED DESCRIPTION:
This is a single arm, multi-institution (1) Hackensack Meridian Health at Hackensack, NJ (2) Jersey Shore Medical Center, Neptune, NJ and (3) Georgetown/Lombardi Cancer Center) phase II study of the combination of pembrolizumab, belantamab, and dexamethasone in patients with triple class refractory multiple myeloma. All institutions will share the same Institutional Review Board.

Safety lead-in Cohort: After the first 10 patients are enrolled, an independent safety review committee will meet to review adverse events and toxicity and determine whether the trial will continue to enroll.

Phase 2 portion: The remainder of patients will be enrolled using a Simon's - 2 stage design.

The study will be conducted in compliance with the International Council for Harmonisation (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use/Good Clinical Practice (GCP) and applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria: Participants are eligible to be included in the study only if all of the following criteria apply:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of multiple myeloma.
2. Patients must have relapsed or must be considered refractory to all of the following:

   1. a proteasome inhibitor,
   2. an immunomodulating agent,
   3. a CD38-monoclonal antibody
   4. an autologous stem cell transplant
   5. CAR T-cell therapy (or ineligible)
3. Patients must have more than 4 lines of prior therapy.
4. Measurable disease, defined as one of the following:

   1. M-protein ≥ 0.5g/dL (0.3 g/dL or above if IgA subtype)
   2. Urine M-protein ≥ 200 mg/24hours
   3. Serum free light chain difference > 100 mg/L
   4. Biopsy proven plasmacytoma
   5. Bone marrow involvement >10%
5. Life expectancy >3 months
6. Eastern Cooperative Oncology Group (ECOG) Performance Score 0-1
7. Adequate hepatic function within 28 days prior to Cycle 1 Day 1 (C1D1):

   1. Total bilirubin < 1.5 × upper limit of normal (ULN) (except patients with Gilbert's syndrome who must have a total bilirubin of < 3 × ULN), and
   2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) normal to <2 × ULN.
8. Adequate renal function within 28 days prior to C1D1 as determined by estimated creatinine clearance of ≥ 30 mL/min, calculated using the Cockcroft and Gault formula (140 - Age) • Mass (kg)/ (72 • creatinine mg/dL); multiply by 0.85 if female (Cockcroft

1976). 9) Adequate hematopoietic function within 7 days prior to C1D1: total white blood cell (WBC) count ≥1500/mm3, absolute neutrophil count ≥1000/mm3, hemoglobin ≥8.5 g/dL and platelet count ≥30,000/mm3 (patients for whom <50% of bone marrow nucleated cells are plasma cells)

a. Patients receiving hematopoietic growth factor support, including erythropoietin, darbepoetin, granulocyte-colony stimulating factor (GCSF), granulocyte macrophage colony stimulating factor (GM-CSF), and platelet stimulators (eg, eltrombopag, romiplostim, or interleukin-11) must have a 2-week interval between growth factor support and the Screening assessments, but they may receive growth factor support during the study. b. Patients must have: i. At least a 2-week interval from the last red blood cell (RBC) transfusion prior to the Screening hemoglobin assessment, and ii. At least a 1-week interval from the last platelet transfusion prior to the Screening platelet assessment. However, patients may receive RBC and/or platelet transfusions as clinically indicated per institutional guidelines during the study. 10) Male and Female Participants: A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 4 months after the last dose of study treatment and refrain from donating sperm during this period. A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 4 months after the last dose of study treatment. -

Exclusion Criteria:

1. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study
2. Any of the following laboratory abnormalities (unless there is >50% plasma cell involvement of the bone marrow):

   1. Absolute neutrophil count (ANC) < 1,000/μL
   2. Platelet count < 30,000/μL
   3. Corrected serum calcium > 13.5 mg/dL (> 3.4 mmol/L)
   4. Serum glutamic oxaloacetic transaminase (SGOT)/aspartate aminotransferase (AST) or serum glutamic pyruvic transaminase (SGPT)/alanine aminotransferase (ALT) ≥ 2.5 x upper limit of normal (ULN)
   5. Serum total bilirubin, direct bilirubin, and alkaline phosphatase ≥ 1.5 x ULNf. Subjects with serious renal impairment ([CrCl] < 50 mL/min) or requiring dialysis would be excluded

   g. International Normalized Ratio (INR) of >1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
3. Subjects with a prior history of malignancies, other than Multiple Myeloma (MM), unless the subject has been free of the disease for ≥ 5 years with the exception of the following noninvasive malignancies:

   1. Basal cell carcinoma of the skin
   2. Squamous cell carcinoma of the skin
   3. Carcinoma in situ of the cervix
   4. Carcinoma in situ of the breast
   5. Incidental histological findings of prostate cancer such as T1a or T1b using the Tumor/Node/Metastasis (TNM) classification of malignant tumors or prostate cancer that is curative
4. Subject has received a prior anti-BCMA therapy
5. Subject has received prior systemic anti-cancer therapy including investigational agents within 3 weeks prior to study intervention
6. Subject has received prior radiotherapy within 2 weeks of start of study intervention.

   Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease
7. Subject has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed
8. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 3 weeks prior to the first dose of study intervention
9. Subject has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
10. Subject has known active Central Nervous System (CNS) metastases and/or carcinomatous meningitis.

    Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 3 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
11. Subject has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
12. Subject has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
13. Subject has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
14. Subject has an active infection requiring systemic therapy.
15. Subject has a known history of Human Immunodeficiency Virus (HIV) infection.

    a. Note: No HIV testing is required unless mandated by local health authority.
16. Subject has active Hepatitis B infection or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis C is required unless mandated by local health authority.
17. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 4 months after the last dose of trial treatment.
18. Subject has had an allogenic tissue/solid organ transplant
19. Subject has uncontrolled ocular disease or keratopathy
20. Subject has uncontrolled cardiovascular disease, specifically uncontrolled hypertension, recent Myocardial Infarction (within 4 months), NYHA Stage 3 or 4 congestive heart failure.
21. Subject is a WOCBP who has a positive urine pregnancy test within 72 hours prior to first dose of study intervention (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
22. Contraindications to the other treatment regimens, as per local prescribing information
23. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 2 years
  To evaluate the overall response rate for pembrolizumab, belantamab and dexamethasone (PBd) in patients with triple class refractory multiple myeloma.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 2 years
  To assess rates of progression-free survival (PFS)
Overall Survival (OS) | 2 years
  To assess rates of overall survival (OS)
Time to next treatment | 2 years
  To assess rates of time to next treatment
Tolerability and Safety | 2 years
  To determine the tolerability and safety of the combination of pembrolizumab with belantamab and dexamethasone by rate of incidence of adverse events using National Cancer Institute (NCI) common terminology criteria for adverse events (CTCAE), v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Noa Biran, MD, Principal Investigator — Division of Hematology and Oncology
Locations (3):
- United States (3):
  - Lombardi Comprehensive Cancer Center, Georgetown University, Washington D.C., District of Columbia
  - John Theurer Cancer Center, Hackensack Meridian Health, Hackensack, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Disis ML. Immune regulation of cancer. J Clin Oncol. 2010 Oct 10;28(29):4531-8. doi: 10.1200/JCO.2009.27.2146. Epub 2010 Jun 1. PMID 20516428
- [Background] Dudley ME, Wunderlich JR, Yang JC, Sherry RM, Topalian SL, Restifo NP, Royal RE, Kammula U, White DE, Mavroukakis SA, Rogers LJ, Gracia GJ, Jones SA, Mangiameli DP, Pelletier MM, Gea-Banacloche J, Robinson MR, Berman DM, Filie AC, Abati A, Rosenberg SA. Adoptive cell transfer therapy following non-myeloablative but lymphodepleting chemotherapy for the treatment of patients with refractory metastatic melanoma. J Clin Oncol. 2005 Apr 1;23(10):2346-57. doi: 10.1200/JCO.2005.00.240. PMID 15800326
- [Background] Hunder NN, Wallen H, Cao J, Hendricks DW, Reilly JZ, Rodmyre R, Jungbluth A, Gnjatic S, Thompson JA, Yee C. Treatment of metastatic melanoma with autologous CD4+ T cells against NY-ESO-1. N Engl J Med. 2008 Jun 19;358(25):2698-703. doi: 10.1056/NEJMoa0800251. PMID 18565862
- [Background] Greenwald RJ, Freeman GJ, Sharpe AH. The B7 family revisited. Annu Rev Immunol. 2005;23:515-48. doi: 10.1146/annurev.immunol.23.021704.115611. PMID 15771580
- [Background] Okazaki T, Maeda A, Nishimura H, Kurosaki T, Honjo T. PD-1 immunoreceptor inhibits B cell receptor-mediated signaling by recruiting src homology 2-domain-containing tyrosine phosphatase 2 to phosphotyrosine. Proc Natl Acad Sci U S A. 2001 Nov 20;98(24):13866-71. doi: 10.1073/pnas.231486598. Epub 2001 Nov 6. PMID 11698646
- [Background] Zhang X, Schwartz JC, Guo X, Bhatia S, Cao E, Lorenz M, Cammer M, Chen L, Zhang ZY, Edidin MA, Nathenson SG, Almo SC. Structural and functional analysis of the costimulatory receptor programmed death-1. Immunity. 2004 Mar;20(3):337-47. doi: 10.1016/s1074-7613(04)00051-2. PMID 15030777
- [Background] Chemnitz JM, Parry RV, Nichols KE, June CH, Riley JL. SHP-1 and SHP-2 associate with immunoreceptor tyrosine-based switch motif of programmed death 1 upon primary human T cell stimulation, but only receptor ligation prevents T cell activation. J Immunol. 2004 Jul 15;173(2):945-54. doi: 10.4049/jimmunol.173.2.945. PMID 15240681
- [Background] Sheppard KA, Fitz LJ, Lee JM, Benander C, George JA, Wooters J, Qiu Y, Jussif JM, Carter LL, Wood CR, Chaudhary D. PD-1 inhibits T-cell receptor induced phosphorylation of the ZAP70/CD3zeta signalosome and downstream signaling to PKCtheta. FEBS Lett. 2004 Sep 10;574(1-3):37-41. doi: 10.1016/j.febslet.2004.07.083. PMID 15358536
- [Background] Riley JL. PD-1 signaling in primary T cells. Immunol Rev. 2009 May;229(1):114-25. doi: 10.1111/j.1600-065X.2009.00767.x. PMID 19426218
- [Background] Parry RV, Chemnitz JM, Frauwirth KA, Lanfranco AR, Braunstein I, Kobayashi SV, Linsley PS, Thompson CB, Riley JL. CTLA-4 and PD-1 receptors inhibit T-cell activation by distinct mechanisms. Mol Cell Biol. 2005 Nov;25(21):9543-53. doi: 10.1128/MCB.25.21.9543-9553.2005. PMID 16227604
- [Background] Francisco LM, Sage PT, Sharpe AH. The PD-1 pathway in tolerance and autoimmunity. Immunol Rev. 2010 Jul;236:219-42. doi: 10.1111/j.1600-065X.2010.00923.x. PMID 20636820
- [Background] Yu B, Jiang T, Liu D. BCMA-targeted immunotherapy for multiple myeloma. J Hematol Oncol. 2020 Sep 17;13(1):125. doi: 10.1186/s13045-020-00962-7. PMID 32943087
- [Background] Raje N, Berdeja J, Lin Y, Siegel D, Jagannath S, Madduri D, Liedtke M, Rosenblatt J, Maus MV, Turka A, Lam LP, Morgan RA, Friedman K, Massaro M, Wang J, Russotti G, Yang Z, Campbell T, Hege K, Petrocca F, Quigley MT, Munshi N, Kochenderfer JN. Anti-BCMA CAR T-Cell Therapy bb2121 in Relapsed or Refractory Multiple Myeloma. N Engl J Med. 2019 May 2;380(18):1726-1737. doi: 10.1056/NEJMoa1817226. PMID 31042825
- [Background] Lonial S, Lee HC, Badros A, Trudel S, Nooka AK, Chari A, Abdallah AO, Callander N, Lendvai N, Sborov D, Suvannasankha A, Weisel K, Karlin L, Libby E, Arnulf B, Facon T, Hulin C, Kortum KM, Rodriguez-Otero P, Usmani SZ, Hari P, Baz R, Quach H, Moreau P, Voorhees PM, Gupta I, Hoos A, Zhi E, Baron J, Piontek T, Lewis E, Jewell RC, Dettman EJ, Popat R, Esposti SD, Opalinska J, Richardson P, Cohen AD. Belantamab mafodotin for relapsed or refractory multiple myeloma (DREAMM-2): a two-arm, randomised, open-label, phase 2 study. Lancet Oncol. 2020 Feb;21(2):207-221. doi: 10.1016/S1470-2045(19)30788-0. Epub 2019 Dec 16. PMID 31859245